CLINICAL TRIAL: NCT07022561
Title: Social Prescribing for Advancing Resilience in Kids (SPARK): A Pilot Study of Social Prescribing for Children and Youth Mental Health in Canada
Brief Title: Social Prescribing for Advancing Resilience in Kids: A Pilot Study of Social Prescribing
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Children's Hospital of Eastern Ontario Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-25-03-0163
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Youth Mental Health and Wellbeing; Feasibility and Acceptability of the Social Prescribing Program
Keywords: social prescribing; children and youth mental health; intervention; wellbeing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social prescribing intervention (Experimental): Youth randomly assigned to the social prescribing intervention group will have access to a social prescribing activity during their 12 weeks of participation.
  Interventions: Behavioral: Social Prescribing
- Educational control (No Intervention): Youth randomly assigned to the educational control will not be provided a social prescribing intervention program, but they will be provided an educational booklet about the importance of connections.

INTERVENTIONS:
Behavioral: Social Prescribing — A social prescribing intervention is a non-clinical approach to improving health and wellbeing by connecting individuals to community-based services and activities that address social, emotional, and practical needs. These may include arts programs, physical activity, peer support, volunteering, or nature-based activities. Facilitated by a link worker or navigator, social prescribing is tailored to the individual and aims to enhance mental health, reduce isolation, and support overall wellness beyond traditional medical care.
  Arms: Social prescribing intervention

SUMMARY:
The goal of this clinical trial is to learn if the Social Prescription (SP) intervention helps improve mental health and wellbeing in youth. It will also assess the feasibility and acceptability of implementing SP in a community setting. The main questions it aims to answer are:

* Is the SP intervention feasible and acceptable for youth, caregivers, and staff?
* Does the SP intervention improve mental health outcomes, reduce stress, and increase wellbeing and social connectedness in youth?

Researchers will compare the Social Prescription (SP) intervention to an education control group to evaluate its effectiveness in improving youth mental health and wellbeing.

Participants will:

* Be randomized to receive either the SP intervention or be placed in an education control group
* Complete wellbeing and mental health questionnaires at the beginning of the study and again after 12 weeks
* Participate in qualitative interviews to share their experiences after participating in SP

ELIGIBILITY:
Inclusion Criteria:

* between 11-17 years of age
* on the waitlist for mental health services
* are not an immediate safety threat to themselves or others as assessed by the HEADS ED questionnaire

Exclusion Criteria:

* Children < 11 years old
* Adolescents > 17 years old

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale | From enrollment to end of treatment or control period at 12 weeks.
  The Revised Children's Anxiety and Depression Scale (RCADS) is a self-report questionnaire that measures symptoms of anxiety and depression in children and adolescents aged 8 to 18.
Perceived Stress Scale | From enrollment to end of treatment or control period at 12 weeks.
  The Perceived Stress Scale is a widely used to help understand how different situations affect our feelings and our perceived stress.
Warwick-Edinburgh Mental Wellbeing Scale | From enrollment to end of treatment or control period at 12 weeks
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) was developed to enable the monitoring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental wellbeing.
Social Connectedness Scale | From enrollment to end of treatment or control period at 12 weeks
  The Social Connectedness Scale measures the extent to which individuals feel connected to others in their social environment.
Student Resilience Survey | From enrollment to end of treatment or control period at 12 weeks
  Student Resilience Survey measuring students' perceptions of their individual characteristics as well as protective factors embedded in the environment:

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | From enrollment to end of treatment or control period at 12 weeks
  The Acceptability of Intervention Measure evaluates how agreeable or satisfactory an intervention is perceived to be by participants or implementers.
Intervention Appropriateness Measure | From enrollment to end of treatment or control period at 12 weeks
  The Intervention Appropriateness Measure assesses the perceived relevance or suitability of an intervention for a specific setting or population.
Feasibility of Intervention Measure | From enrollment to end of treatment or control period at 12 weeks
  The Feasibility of Intervention Measure gauges how practical and possible it is to implement an intervention within a given setting.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Racine, PhD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data outside of our affiliations and institutions.

REFERENCES:
- [Derived] Kempe S, Bennett S, MacLeod O, Mohamed N, Cloutier P, Muhl C, Hayes D, Mitsakakis N, Goldfield G, Racine N. Social prescriptions for advancing resilience in kids (SPARK): study protocol for a randomized controlled trial. BMC Psychol. 2025 Oct 10;13(1):1126. doi: 10.1186/s40359-025-03465-7. PMID 41074116